CLINICAL TRIAL: NCT05043467
Title: Retrospective Study to Evaluate the Safety of Duvie in Korean Patients With Type 2 Diabetes Mellitus
Acronym: DISCOVERY
Status: Completed | Type: Observational
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 59DM17022
Record Dates: First submitted 2021-09-03; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duvie(Lobeglitazone): patients with type 2 diabetes who received lobeglitazone 0.5mg for more than one year between February 1, 2014 and December 20, 2018
  Interventions: Drug: Duvie(Lobeglitazone) tab 0.5mg

INTERVENTIONS:
Drug: Duvie(Lobeglitazone) tab 0.5mg — patients with type 2 diabetes who received lobeglitazone 0.5mg for more than one year between February 1, 2014 and December 20, 2018
  Other Names: Chong Kun Dang Pharmaceutical, Duvie tab 0.5mg, code no.(643306610)

SUMMARY:
Previous thiazolidinediones (TZDs) have issued various safety concerns including weight gain, bladder cancer, and congestive heart failure (CHF). This study aimed to evaluate the efficacy and safety of lobeglitazone, a novel TZD in patients with type 2 diabetes in real world.

DETAILED DESCRIPTION:
Lobeglitazone have clinical trials conducted in Korean type 2 diabetics patients for 6 months to up to 12 months, and the results of study on the efficacy and safety of lobeglitazone are relatively limited. In pre-marketing clinical trials, a controlled group of patients is enrolled to minimize other possible effects in determining the efficacy and safety of the drug.

Consequently, in real clinical practice, unexpectable safety information that has not been discovered at the pre-marketing stage may accur because it is more extensively and longer administered to a variety of patients who may have various underlying conditions and diseases. Therefore, there should be an ongoing assessment of safety information in real world. There have been the safety concerns of TZD, such as congestive heart failure (CHF), fractures, bladder cancer (long-term use), edema, and weight gain. Previous study has reported that lobeglitazone has better safety on bladder cancers and bone fractures than other TZDs, but currently, there is a lack of large-scaled, long-term safety and efficacy data of lobeglitazone in Korean real practice.

This is a non-interventional, multi-centered, retrospective and observational study and aimed to evaluate the efficacy and safety of lobeglitazone in patients with type 2 diabetes in real world.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes who received lobeglitazone 0.5mg for more than one year between February 1, 2014 and December 20, 2018

Exclusion Criteria:

* patients who are not appropriate to participate in this research based on principal investigators' decision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who satisfy the inlusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 2228 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Incidence of major adverse events (AEs) and any AEs that occurred during the administration period of lobeglitazone | during the administration period of lobeglitazone
  Investigators identified the following as major AEs: edema, weight gain(in kilograms), fractures, bladder cancer, anemia, hypoglycemia, macular edema, cardiac death, myocardial Infarction, stroke, transient ischemic attack, coronary arterial occlusion, and CHF. Investigators also identified any AEs including blood pressure(in millimeter of mercury) change, increased liver enzyme (> 3X), and dizziness.

SECONDARY OUTCOMES:
Changes in glycated hemoglobin (HbA1c) and glucose, lipid parameters | 3, 6, 12, 18, 24, 36, 42, and 48 months after administration of lobeglitazone
  Investigators identified changes in glycated hemoglobin (HbA1c in percentage) and glucose(in milligrams per deciliter), lipid parameters in milligrams per deciliter(total cholesterol, triglyceride, low-density lipoprotein [LDL] cholesterol, and high-density lipoprotein [HDL] cholesterol) at 3, 6, 12, 18, 24, 36, 42, and 48 months after administration of lobeglitazone.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Rae S Kim, M.D, PhD, Principal Investigator — Division of Endocrinology and Metabolism, Department of Internal Medicine, Bucheon St Mary's Hospital
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Bucheon St Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No